CLINICAL TRIAL: NCT04883944
Title: Maternal Involvement in Pain Management in NICU: a Randomized Controlled Trial
Brief Title: Maternal Involvement in Pain Management in NICU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: Co.Ma.Do./2021
Record Dates: First submitted 2021-05-07; First posted 2021-05-12 (Actual); Last update posted 2022-05-23 (Actual); Status verified 2022-05

CONDITIONS: Procedural Pain; Mother-Infant Interaction; Infant, Newborn; Stress, Physiological
Keywords: NICU, newborn, pain, Parental stress, nurse
MeSH Terms: conditions — Pain, Procedural; Pain

STUDY DESIGN:
Intervention Model Description: a prospective, randomized controlled trial with a 2x2 crossover design
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): All the enrolled infants will receive the heel stick procedure with the maternal involvement after mother will be trained on the application of the non-pharmacological techniques during the performance of the procedure.
  Interventions: Other: Intervention group
- Standard care (Active Comparator): All the enrolled infants will receive the heel stick procedure according to local protocol without the maternal involvement. The non-pharmacological techniques will be performed by a second nurse not involved in the heel stick procedure itself.
  Interventions: Other: Standard care group

INTERVENTIONS:
Other: Intervention group — Mother will be involved in implementing the non-pharmacological techniques during the performance of the heel stick procedure as follow:
  * swaddling;
  * non-nutritive sucking with pacifier in infants with PMA < 32 weeks;
  * nutritional sucking with sucrose and/or breast milk in infants with PMA ≥ 32 weeks;
  * holding;
  * exposure to maternal voice.
  Arms: Intervention group
Other: Standard care group — A second nurse will perform the non-pharmacological techniques during the performance of the heel stick procedure without the maternal involvement as follow:
  * swaddling;
  * non-nutritive sucking with pacifier in infants with PMA < 32 weeks;
  * nutritional sucking with sucrose and/or breast milk in infants with PMA ≥ 32 weeks;
  * holding.
  Arms: Standard care

SUMMARY:
Infants admitted to Neonatal Intensive Care Unit (NICU) may experience a negative impact due to multiple painful and stressful procedures during their hospitalization. The American Academy of Pediatrics recommends that healthcare facilities taking care of newborns should implement pain prevention and management programs.

There are some non-pharmacological techniques that have been developed to reduce newborn's pain perception, including swaddling, holding, non-nutritive sucking in infants with Post-menstrual age (PMA) below 32 weeks, nutritional sucking with the administration of breast milk or sweeteners above 32 weeks PMA and exposure to maternal voice.

Even for parents, the experience of NICU hospitalization of their child is a particularly stressful event, mainly characterized by feelings of exclusion due to lack of interactions with their own baby due to their clinical conditions.

Hence, it is very important to intervene as soon as possible on parental stress that can affect the physical and psychological quality of life of the family. This is possible through the application of nursing care plans that involve the parents in daily care and support them in the long process of development and acquisition of autonomy and skills.

The nurse is a healthcare provider who has the most frequent contact with newborns hospitalized in NICU and has a key role in preventing, recognizing, and managing newborn's pain. However, there is a considerable discrepancy between the theory and practice: many nurses and doctors are aware that most of the procedures carried out in NICU cause pain.

Therefore, nurses also can develop high levels of physical and psychological stress, particularly when they manage a newborn who feels pain.

The purpose of this study is to evaluate if maternal involvement in the pain management of newborn admitted to NICU may reduce the level of pain perceived by infant during the heel stick procedure using the Premature Infant Pain Profile (PIPP) pain scoring tool. In addition, the study's secondary goal will be to investigate if maternal involvement in pain management of newborn may produce positive effects on the mother in reducing stress, depression and anxiety and in reducing nurses' physical and psychological stress.

DETAILED DESCRIPTION:
This study is a prospective, randomized controlled trial with a 2x2 crossover design. Study population include newborns admitted to NICU that require a heel stick procedure after the first week of life, mothers of enrolled infants and nurses performing the heel stick procedure. The sample size will be 50 newborns who meet the inclusion criteria. Newborns will be randomly assigned to receive: i) a heel stick procedure with maternal involvement and after a week an heel stick procedure without maternal involvement or ii) a procedure without maternal involvement and after a week a procedure with maternal involvement. For both group the washout period between the two procedures is 7 days.

Before the intervention with the maternal involvement, mother will receive a training regarding the heel stick procedure and pain management.

Research hypothesis:

H1. Newborns receiving the intervention with the maternal involvement during the heel stick procedure have lower pain level than those who receive the intervention without the maternal involvement.

H2. Mothers who are involved in their baby pain management during the heel stick procedure have lower level of stress, anxiety and depression than those who are not involved during the painful procedure.

H3. Nurses have a positive effect in term of reducing stress level if mother is involved in pain management of own baby.

PIPP (Premature Infant Pain Profile) scale will be used to evaluate the pain response during the heel stick procedure. The level of stress, anxiety and depression of mother and the stress level of nurse will be assessed with validated questionnaires.

ELIGIBILITY:
Inclusion Criteria:

For infants:

- Infants born ≥ 23 weeks of gestational age who require an heel stick procedure, after the first week of life

For mothers:

- Mothers' age over 18 years and good comprehension of Italian language

For nurses:

- Nurses or pediatric nurses with professional experience in NICU ≥ 6 months who decide to participate at the study

Exclusion Criteria:

For infants:

* Enteral and/or parenteral sedation/analgesia ongoing or suspended less than 4 hours from the beginning of the procedure
* Infants who receive multiple painful procedures at the same time

For mothers:

* bad comprehension of Italian language
* age under 18 years

For nurses:

* Nurses and pediatric nurses with professional experience in NICU ≤ 6 months
* Nurses and pediatric nurses who don't give consent to study participation

Ages: 1 Week to 1 Month | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2021-05-17 (Actual); Primary Completion 2022-05-16 (Actual); Study Completion 2022-05-16 (Actual)

PRIMARY OUTCOMES:
Newborn's pain response during the performance of the heel stick procedure | From 15 seconds before heel stick to 30 seconds after the end of the procedure
  Pain score calculated with the Premature Infant Pain Profile (PIPP) pain scoring tool one time for each procedure. The scale require an observation starting 15 seconds before the heel stick to 30 seconds after the end of the procedure. This score varies from "0" (no pain) to "21" (maximun pain response).

SECONDARY OUTCOMES:
Anxiety, stress and depression of mother | From the date of inclusion until the date of completion study, measured up to 15 days
  Mean scores of maternal stress of infants enrolled will be evaluated with the Parental Stressor Scale - NICU and Depression, Anxiety and Stress Scale, measured at the beginning of the study and after having performed each heel stick procedure, in both arms of study.
Stress levels of nurse performing heel stick | From the date of inclusion until the date of completion study, measured up to 15 days
  Mean score of stress level of nurse who performs the heel stick will be evaluated with the Rapid stress assessment scale (an Italian validated scale), measured at the beginning of the study and after having performed each heel stick procedure, in both arms of study.

CONTACTS AND LOCATIONS:
Overall Officials: Agostino Guarino, RN, Principal Investigator — Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico
Locations (1):
- Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico, NICU, Milan, MI, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] COMMITTEE ON FETUS AND NEWBORN and SECTION ON ANESTHESIOLOGY AND PAIN MEDICINE. Prevention and Management of Procedural Pain in the Neonate: An Update. Pediatrics. 2016 Feb;137(2):e20154271. doi: 10.1542/peds.2015-4271. Epub 2016 Jan 25. PMID 26810788
- [Background] Axelin A, Lehtonen L, Pelander T, Salantera S. Mothers' different styles of involvement in preterm infant pain care. J Obstet Gynecol Neonatal Nurs. 2010 Jul-Aug;39(4):415-24. doi: 10.1111/j.1552-6909.2010.01150.x. PMID 20629928
- [Background] Bellieni CV, Buonocore G, Nenci A, Franci N, Cordelli DM, Bagnoli F. Sensorial saturation: an effective analgesic tool for heel-prick in preterm infants: a prospective randomized trial. Biol Neonate. 2001 Jul;80(1):15-8. doi: 10.1159/000047113. PMID 11474143
- [Background] Bottesi G, Ghisi M, Altoe G, Conforti E, Melli G, Sica C. The Italian version of the Depression Anxiety Stress Scales-21: Factor structure and psychometric properties on community and clinical samples. Compr Psychiatry. 2015 Jul;60:170-81. doi: 10.1016/j.comppsych.2015.04.005. Epub 2015 Apr 15. PMID 25933937
- [Background] Busse M, Stromgren K, Thorngate L, Thomas KA. Parents' responses to stress in the neonatal intensive care unit. Crit Care Nurse. 2013 Aug;33(4):52-9; quiz 60. doi: 10.4037/ccn2013715. PMID 23908169
- [Background] Cruz MD, Fernandes AM, Oliveira CR. Epidemiology of painful procedures performed in neonates: A systematic review of observational studies. Eur J Pain. 2016 Apr;20(4):489-98. doi: 10.1002/ejp.757. Epub 2015 Jul 29. PMID 26223408
- [Background] Lago P, Garetti E, Merazzi D, Pieragostini L, Ancora G, Pirelli A, Bellieni CV; Pain Study Group of the Italian Society of Neonatology. Guidelines for procedural pain in the newborn. Acta Paediatr. 2009 Jun;98(6):932-9. doi: 10.1111/j.1651-2227.2009.01291.x. PMID 19484828
- [Background] Lovibond PF, Lovibond SH. The structure of negative emotional states: comparison of the Depression Anxiety Stress Scales (DASS) with the Beck Depression and Anxiety Inventories. Behav Res Ther. 1995 Mar;33(3):335-43. doi: 10.1016/0005-7967(94)00075-u. PMID 7726811
- [Background] Miles MS, Funk SG, Carlson J. Parental Stressor Scale: neonatal intensive care unit. Nurs Res. 1993 May-Jun;42(3):148-52. PMID 8506163